CLINICAL TRIAL: NCT03478657
Title: An Open-label Study to Evaluate Correct Use and Ease of Use of the ELLIPTA Dry Powder Inhaler (DPI) in Pediatric Patients Currently Receiving Inhaled Therapy for Treatment of Their Asthma
Brief Title: An Open-label Study to Evaluate Correct Use and Ease of Use of the ELLIPTA DPI in Pediatric Subjects With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 206924
Record Dates: First submitted 2018-03-22; First posted 2018-03-27 (Actual); Results first posted 2019-12-09 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-02

CONDITIONS: Asthma
Keywords: Asthma; Dry Powder Inhaler; Metered Dose Inhaler; Long Acting beta 2 Agonist; ELLIPTA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Subjects from the age group of 5 to 11 years with documented history of symptoms of asthma or diagnosis of asthma for at least 6 months prior to Visit 1 will be assessed for the ease of use of ELLIPTA DPI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects using placebo ELLIPTA DPI (Experimental): Subjects in stratum 1 and stratum 2 will be of age group from 5 to 7 years and 8 to 11 years respectively. Subjects will take placebo ELLIPTA DPI once daily. During Visit 2 (Day 28) subjects will be randomized to receive questionnaire on ELLIPTA DPI usage either version A or B.
  Interventions: Drug: Placebo DPI; Device: ELLIPTA DPI; Other: Ease of use questionnaires

INTERVENTIONS:
Drug: Placebo DPI — Subjects will receive placebo via oral inhalation route using ELLIPTA once daily. Placebo DPI will be available in two strips of 30 blisters per strip. First strip will contain lactose monohydrate and second strip will have lactose monohydrate blended with magnesium stearate.
Device: ELLIPTA DPI — Subjects will receive placebo DPI via ELLIPTA. ELLIPTA is trademark of GSK
Other: Ease of use questionnaires — Subjects from both stratum after use of ELLIPTA DPI will be randomized to receive either version A or B of the questionnaires. Subjects will be asked questions on ease of use of ELLIPTA. Parent/guardian will also complete a questionnaire about the ELLIPTA DPI.

SUMMARY:
Asthma is a chronic inflammatory disease of airways and lungs that results in hyper-reactivity and clinically relevant episodes of wheezing. This study has been designed to assess the correct use and ease of use of the ELLIPTA® DPI in pediatric subjects with asthma. ELLIPTA DPI is easy to use, requires few steps, is consistent in dosing and eliminates the hand-breath co-ordination required for metered dose inhalers (MDIs). Subjects will be stratified by age into two strata: Stratum 1: subjects in the age group of 5 to 7 years and Stratum 2: Subjects in the age group of 8 to 11 years. All subjects will be trained by Health care professionals (HCP) for the correct use of ELLIPTA DPI. Subjects will be given three chances to attempt correct use of ELLIPTA DPI; subsequently, if the subject is not successful, the parent/guardian will be able to help instruct the subject on the correct use of the ELLIPTA DPI, for two more attempts. The subjects who will be enrolled in the study will take placebo ELLIPTA DPI once daily. After 28 days subjects will be randomized in 1:1 to receive a questionnaire (Version A and B). After completion of the questionnaire on ELLIPTA DPI ease of use, subject's ability to use ELLIPTA DPI correctly will be re-assessed. Approximately 219 subjects will be screened to participate in the study. The study will be conducted for 28 days. ELLIPTA is a registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 5 and 11 years old (inclusive), at the time of the Visit 0.
* Subjects with a documented history of symptoms consistent with a diagnosis of asthma for at least 6 months prior to V0 (includes asthma diagnosis).
* Males and premenarchial females.
* Written informed consent from at least one parent/guardian and the accompanying informed assent from the subject (where the subject is able to provide assent) prior to admission to the study.
* Subject and their legal guardian understand and are willing, able, and likely to comply with study procedures and assessments.
* Subject must have been receiving asthma treatment (rescue or maintenance) for 3 months prior to entry onto the study.
* Subject must have never been trained in correct use of, or used the ELLIPTA DPI previously.
* Subjects must be able to demonstrate correct use of the ELLIPTA DPI after coaching/training at Visit 1.
* Subjects must be able to converse and understand verbal instruction in English.

Exclusion Criteria:

* Subjects with concurrent diagnosis of other respiratory disorders including active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases, cystic fibrosis or other active pulmonary diseases.
* Subjects with concurrent diagnosis of psychiatric or psychological or any other disorders that in the opinion of the investigator may affect the ability of the subject to comply with study procedures or requirements.
* Subject has experienced an exacerbation which required oral/systemic corticosteroids in the three months prior to Visit 0.
* Subject has been hospitalized for an episode of asthma within three months of Visit 0.
* Subject has had an asthmatic episode requiring intubation, associated with hypercapnia, respiratory arrest or hypoxic seizures.
* Subject has exhibited symptoms of a recent acute respiratory tract infection within one week of Visit 0.
* Subject has history of hypersensitivity to any components of the study inhalers (example [e.g.], lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation will also be excluded.
* Subjects with historical or current evidence of clinically significant or rapidly progressing or unstable cardiovascular, neurological, renal, hepatic, immunological, endocrine (including diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the analysis if the disease/condition exacerbated during the study.
* Parent or Guardian with a history of psychiatric disease, intellectual deficiency, substance abuse or other condition (e.g. inability to read, comprehend or write) which may affect: Validity of consent to participate in the study; Adequate supervision of the subject during the study; Compliance of subject with study medication and study procedures; subject safety and well-being.
* Subjects who have received an investigational drug and/or medical device within 30 days of entry into this study (Screening), or within five drug half-lives of the investigational drug, whichever is longer.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (19):
- United States (15):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Napa, California
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Waco, Texas
- Canada (4):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20765

REFERENCES:
- [Derived] Halverson P, Liem J, Heyes L, Preece A, Bareille P, Rees J, Jain R, Stanford RH, Lenney W, Collison K, Sharma R. The evaluation of the correct use and ease-of use of the ELLIPTA DPI in children with asthma. Pediatr Pulmonol. 2021 Jan;56(1):57-64. doi: 10.1002/ppul.25149. Epub 2020 Nov 19. PMID 33124762
- See also: 206924 Full Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=206924&attachmentIdentifier=b4321234-3409-4cf7-b77d-c77242ab6a9f&fileName=gsk-206924-protocol-redact.pdf&versionIdentifier=
- See also: 206924 Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217381&parentIdentifier=206924&attachmentIdentifier=f5465b2a-409b-445e-bc96-fe3671501308&fileName=gsk-206924-reporting-and-analysis-plan-redact.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, single arm, stratified, open-label, randomized placebo-only study conducted in pediatric participants. Participants were stratified based on age at Visit 0 (Stratum 1: 5 to 7 years old inclusive and Stratum 2: 8 to 11 years old inclusive).
Pre-assignment Details: A total of 232 participants were screened, of which 10 failed screening and 222 participants were enrolled in the study. The study was conducted in the United States and Canada.
Groups:
- Stratum 1: 5-7 Years: Participants received an oral inhalation of placebo once daily via ELLIPTA dry powder inhaler (DPI) for 28 days. At Day 28 (Visit 2), participants received a questionnaire on ease of use of ELLIPTA DPI. Participants were asked questions on ease of use and asked to perform correct use of the ELLIPTA DPI.
- Stratum 2: 8-11 Years: Participants received an oral inhalation of placebo once daily via ELLIPTA DPI for 28 days. At Day 28 (Visit 2), participants received a questionnaire on ease of use of ELLIPTA DPI. Participants were asked questions on ease of use and asked to perform correct use of the ELLIPTA DPI
Period: Overall Study
Arm/Group | Stratum 1: 5-7 Years | Stratum 2: 8-11 Years
Started | 88 | 134
Completed | 88 | 133
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1: 5-7 Years | Stratum 2: 8-11 Years | Total
Number analyzed (Participants) | 88 | 134 | 222
Age, Continuous [Mean (Standard Deviation); unit: Years] — The Intent-to-Treat (ITT) population consists of all participants who have been screened and received at least one dose of the study medication (placebo)
  Years | 6.1 (0.80) | 9.7 (1.10) | 8.3 (2.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 89
  Male | 47 | 86 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Central/South Asian Heritage | 5 | 11 | 16
  Asian-Japanese Heritage | 0 | 1 | 1
  Asian-South East Asian Heritage | 2 | 1 | 3
  Black Or African American | 24 | 37 | 61
  White-Arabic/North African Heritage | 4 | 1 | 5
  White-White/Caucasian/European Heritage | 49 | 75 | 124
  Multiple | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants From Each Stratum Who Demonstrated Correct Use of the ELLIPTA DPI at Visit 2, Attempt 1 (Day 28)
Description: Participants were trained in the correct use of ELLIPTA DPI by a healthcare professional (HCP) on Day 1 (Visit 1) following which eligible participants were required to take one inhalation of placebo from the ELLIPTA DPI once daily for 28 days. At Day 28 (Visit 2), participants were administered a questionnaire on ease of use of ELLIPTA DPI. Participants and their parents/guardian were required to complete the questionnaire, following which participants were assessed for their ability to demonstrate correct use of ELLIPTA DPI (1 attempt with no training or instruction and then 1 attempt after instruction from parent/guardian). Percentage of participants who demonstrated correct use of ELLIPTA was calculated as "number of participants who demonstrated correct use at Visit 2" divided by "number of participants whose use of the ELLIPTA DPI was evaluated at Visit 2" multiplied by 100. The 95% confidence interval (CI) was calculated using the exact binomial distribution.
Time Frame: At Day 28
Population: Modified intent to treat (MITT) Population comprised of all participants who were screened, received at least one dose of the study medication (placebo) and were randomized to a version of the ease of use questionnaire at Visit 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum 1: 5-7 Years | Stratum 2: 8-11 Years
Number analyzed (Participants) | 88 | 133
Percentage of participants | 92 [84 to 97] | 93 [88 to 97]

2. Primary Outcome: Percentage of Participants Who Rated the ELLIPTA DPI as Easy to Use Among Those Who Could Demonstrate Correct Use at Visit 2, Attempt 1 (Day 28)
Description: Participants were trained in the correct use of ELLIPTA DPI at Visit 1 by the HCP and eligible participants were required to take one inhalation of placebo from the ELLIPTA DPI once daily for 28 days. At Day 28 (Visit 2), participants were administered a questionnaire on the ease of use of ELLIPTA DPI. For participants in Stratum 1, questionnaire was provided to the interviewer and responses were recorded. For Stratum 2, the questionnaire was self-administered (or interviewer administered, if participant was unable to self-administer). Percentage of participants who rated the ELLIPTA DPI as easy to use was calculated as "number of participants who rate the ELLIPTA as easy" divided by "number of participants who demonstrated correct use at Visit 2 (Attempt #1)" multiplied by 100. The 95% CI for the percentages are calculated using the exact binomial distribution.
Time Frame: At Day 28
Population: MITT Population. Only those participants who demostrated correct use at Visit 2, attempt 1 has been analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum 1: 5-7 Years | Stratum 2: 8-11 Years
Number analyzed (Participants) | 81 | 124
Percentage of participants | 98 [91 to 99] | 98 [93 to 99]

3. Secondary Outcome: Percentage of Participants From Each Stratum Who Demonstrated Correct Use of the ELLIPTA DPI at Visit 1, Attempt 1 (Day 1)
Description: Participants were trained by HCP in correct use of ELLIPTA DPI at Visit 1 following which participants were assessed on their ability to use the ELLIPTA DPI without guidance from the HCP or parent/guardian. The participants were given a maximum of five attempts. Participants who were unable to use the ELLIPTA DPI correctly were trained by the HCP for the first three attempts. For the fourth and fifth attempts, the participants' parent/guardian assisted in the training of the ELLIPTA DPI. Percentage number of participants who demonstrated correct use of the ELLIPTA DPI along with 95% CI at Visit 1 (attempts 1 to 5) has been presented. The 95% CI for the percentages are calculated using the exact binomial distribution.
Time Frame: Day 1
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum 1: 5-7 Years | Stratum 2: 8-11 Years
Number analyzed (Participants) | 88 | 134
Percentage of participants | 24 [15 to 34] | 50 [41 to 59]

4. Secondary Outcome: Percentage of Participants Who Demonstrated Correct Use of the ELLIPTA DPI at Visit 2, Attempt 1 in All Participants (Stratum 1+Stratum 2)
Description: Participants were trained in the correct use of ELLIPTA DPI by a HCP on Day 1 (Visit 1) following which eligible participants were required to take one inhalation of placebo from the ELLIPTA DPI once daily for 28 days. At Day 28 (Visit 2), participants were administered a questionnaire on ease of use of ELLIPTA DPI. Participants and their parents/guardian were required to complete the questionnaire, following which participants were assessed for their ability to demonstrate correct use of ELLIPTA DPI (1 attempt with no training or instruction and then 1 attempt after instruction from parent/guardian). Percentage of participants who demonstrated correct use of ELLIPTA was calculated as "number of participants who demonstrated correct use at Visit 2" divided by "number of participants whose use of the ELLIPTA DPI was evaluated at Visit 2" multiplied by 100. The 95% CI was calculated using the exact binomial distribution.
Time Frame: At Day 28
Population: MITT Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Stratum 1 + Stratum 2: All participants from Stratum 1 and Stratum 2 (5 to 11 years) were included.
Arm/Group | Stratum 1 + Stratum 2
Number analyzed (Participants) | 221
Percentage of participants | 93 [89 to 96]

5. Secondary Outcome: Percentage of Participants Who Rated Easy Use of ELLIPTA DPI at Visit 2 in All Participants (Stratum 1+Stratum 2)
Description: as for outcome 2
Time Frame: At Day 28
Population: MITT Population. Only those participants who demonstrated correct use at Visit 2, attempt 1 were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum 1 + Stratum 2
Number analyzed (Participants) | 205
Percentage of participants | 98 [94 to 99]

6. Secondary Outcome: Percentage of Participants Who Reported at Least One Critical Error From Each Stratum With the Use of ELLIPTA DPI at Visit 1, Attempt 1
Description: Participants were trained by HCP in correct use of ELLIPTA DPI at Visit 1 following which participants were assessed on their ability to use the ELLIPTA DPI without guidance from the HCP or parent/guardian. The participants were given a maximum of five attempts. Participants who were unable to use the ELLIPTA DPI correctly were trained by the HCP for the first three attempts. For the fourth and fifth attempts, the participants' parent/guardian assisted in the training of the ELLIPTA DPI. Percentage of participants who has withdrawn at any point throughout the correct use demonstration and performed a critical error, was considered as one who performed at least one critical error. Participant who has withdrawn at any point throughout correct use demonstration and did not perform all the critical error items were also considered as one who performed at least one critical error. The 95% CI for the percentages are calculated using the exact binomial distribution.
Time Frame: Day 1
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Stratum 1: 5-7 Years | Stratum 2: 8-11 Years
Number analyzed (Participants) | 88 | 134
Percentage of participants | 51 [40 to 62] | 25 [18 to 34]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected up to Day 28
Description: SAEs and non-SAEs were summarized for the ITT Population. Since all participants received placebo as treatment, data has been combined for all the arms.
Arm/Group | Stratum 1 + Stratum 2
All-Cause Mortality (participants affected / at risk) | 0/222
Serious Adverse Events (participants affected / at risk) | 0/222
Other Adverse Events (participants affected / at risk) | 11/222
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 + Stratum 2 (N=222)
Viral upper respiratory tract infection (Infections and infestations) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT03478657/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT03478657/SAP_001.pdf